CLINICAL TRIAL: NCT05579678
Title: APOLLO: Personalized rehAbilitation PrOgram in aLLOgeneic Bone Marrow Transplantation
Acronym: APOLLO
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA.CC-22-0164
Record Dates: First submitted 2022-09-20; First posted 2022-10-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Allogeneic Disease
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Supportive nursing, nutritional and physical activity with a handheld 'app' — Supportive nursing, nutritional and physical activity with a handheld 'app'

SUMMARY:
People who undergo allogeneic bone marrow transplant for blood cancers receive the highest chemotherapy doses possible that humans can receive and still survive. As a result, they have devastating side effects during the procedure and for many years afterwards. Damage to organs and muscles cause long-lasting physical weakness and the psychological experience is severe enough to be termed 'post traumatic stress disorder' that also lasts for many years. These effects are worsened by the fact that most Canadians live several hours away from treatment and transplant centers, leaving them entirely on their own to manage these difficult long term effects. The APOLLO team will perform a qualitative study to learn the experiences of people undergoing allogeneic bone marrow transplant while they receive access to a supportive care computer 'app' and telephone support from nursing, exercise and nutrition experts. In this way, the APOLLO team will learn the most helpful type and timing of supportive care from those who know best.

ELIGIBILITY:
Inclusion Criteria:

* eligible for allogeneic transplantation

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals scheduled to undergo allogeneic transplantation
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Title: Acceptability of a multimodal supportive care | 1 year
  Description: Questionnaire to assess usefulness of a multimodal supportive care App that includes care navigation (nursing, exercise, nutrition)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pituskin E, Foulkes S, Skow RJ, McMurtry T, Kruger C, Bates JE, Lamoureux D, Brandwein J, Lieuw E, Wu C, Zhu N, Wang P, Sawler D, Taparia M, Hamilton M, Comfort-Riddle T, Meyer T, Gyenes GT, Paterson I, Prado CM, Haykowsky MJ, Greiner JG, McNeely ML, Tandon P, Thompson RB. Rationale and design of APOLLO: a personalized rehAbilitation PrOgram in aLLOgeneic bone marrow transplantation. BMC Cancer. 2025 Jan 28;25(1):163. doi: 10.1186/s12885-025-13502-8. PMID 39875816